CLINICAL TRIAL: NCT03849547
Title: Development of a Smartphone-based System for Training Subjects With Chronic Ankle Instability and Training Effect Evaluation
Brief Title: Evaluation for the Effect of Smartphone Based Training on Chronic Ankle Instability Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Wen-Hsu Sung, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAItraining
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Chronic Ankle Instability
Keywords: Chronic ankle instability; Smartphone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- App training group (Experimental): Subjects in App training group will receive App Balance training via smartphone application.
  Interventions: Other: App Balance training
- Home training group (Active Comparator): Subjects in Home training group will receive Home Balance training advised by physical therapist.
  Interventions: Other: Home Balance training
- Control group (No Intervention): Control group will receive only education of ankle injury prevention related information.

INTERVENTIONS:
Other: App Balance training — Training specially designed for balance ability of chronic ankle instability groups.
  Guidance through smartphone application as home program.
  Arms: App training group
Other: Home Balance training — Training specially designed for balance ability of chronic ankle instability groups.
  Follow the usual home program provided in clinics.
  Arms: Home training group

SUMMARY:
This study aims to verify the training effect of smartphone-based training for chronic ankle instability(CAI) subjects. By randomizing subjects to App training group, clinical training group and control group, the training effect will be compared among groups.

DETAILED DESCRIPTION:
Postural control ability may be damaged after ankle sprains. Poor postural control ability is the risk factors of the ankle sprain, forming a vicious circle of recurrent sprains. Proper and early assessment is the key to breaking down the circle. Smartphones have been utilized in the medical field. With built-in sensors, utilizing smartphones as assessment tools can provide quantitative data of postural control performance. This study aims to verify the training effect of smartphone-based training for CAI subjects.

CAI subjects were recruited and randomly assigned to App training group, Home training group and control group, receiving 6 weeks of intervention. Pre-test was conducted before the intervention, and the post-test was conducted after the 6-week intervention. The follow up assessment was conducted 4 weeks after the post-test.

ELIGIBILITY:
Inclusion Criteria:

* At least one ankle sprain history
* At least 2 times of sprain and feeling unstable
* Diagnosed as functional ankle instability
* Full recovered from injury
* Cumberland Ankle Instability Tool<24
* Ankle Instability Instrument >5 yes
* Identification of Functional Ankle Instability >11

Exclusion Criteria:

* Diagnosis as mechanical instability
* Neurological deficits
* Lower extremity injury within the past 6 wk
* History of lower-extremity surgery
* Other conditions known to affect balance

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Postural sway measurement | 30 seconds
  Using smartphone application and force plate to record the postural sway during single leg stance.
Star Excursion Balance Test | 5 minutes
  To assess the dynamic balance ability of subjects.

SECONDARY OUTCOMES:
Foot and Ankle Outcome Score | 5 minutes
  An ankle function assessment tool, with 5 dimensions includes symptoms, pain, activity, function and sport, and quality of life.
  The scale score ranges from 0% to 100%, the higher the percentage, the better ankle function. Subjects answer the questions by choosing different choices that describe their condition the best.
  The total score will be summed up and calculated as percentage.
Foot and Ankle Ability Measure-sport subscale | 5 minutes
  An ankle function assessment tool. The scale score ranges from 0% to 100%, the higher the percentage, the better ankle function. Subjects answer the 7 questions by choosing different degree of difficulty to accomplish the activities.
  The total score will be summed up and calculated as percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Hsu Sung, Dr., Study Chair — National Yang Ming Chiao Tung University
Locations (1):
- Yang Ming university, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No